CLINICAL TRIAL: NCT02222961
Title: A Single-blind, Placebo-controlled Single Increasing Dose Tolerance Study in Healthy Male Volunteers After Intravenous Administration of BIIR 561 CL as Loading Dose (Dosage: 37.5 mg/h - 150 mg/h, Infusion Time 1 Hour) Followed by Maintenance Dose (Dosage: 20 mg/h - 40 to 125 mg/h), Infusion Time 5 Hours
Brief Title: Single Increasing Dose Followed by Maintenance Dose Tolerance Study of BIIR 561 CL in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 600.2
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — irampanel

ARMS (2):
- BIIR 561 CL (Experimental)
  Interventions: Drug: BIIR 561 CL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIR 561 CL
  Arms: BIIR 561 CL
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of the present study is to obtain information about the safety, tolerability and pharmacokinetics of BIIR 561 after continuous intravenous administration of increasing doses in healthy young volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Age 21 to 50 years
* Broca index from -20% to +20%
* Written informed consent prior to admission to the study

Exclusion Criteria:

* Medical examination, laboratory tests or ECG judged by the investigator to differ significantly from normal clinical values
* Known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Known diseases of the central nervous system (CNS) (such as epilepsy), CNS trauma in their medical history or with psychiatric or neurological disorders
* Known history of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* Allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of a drug with a long half-life (> 24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study
* Intake of any other drug which might influence the results of the trial during the week previous to the start of the study
* Participation in another study with an investigational drug within the last two months preceding this study
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Alcohol use of more than 60 g per day
* Drug dependency
* Excessive physical activities (e.g. competitive sports) within the last week before the study
* Blood donation within the last 4 weeks (>= 100 ml)

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Start 1999-11; Primary Completion 2000-06 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | up to 8 days after drug administration
Number of subjects with clinically significant findings in vital functions | up to 8 days after drug administration
  blood pressure, pulse rate, respiratory rate, oral body temperature
Number of subjects with clinically significant findings in ECG | up to 8 days after drug administration
Number of subjects with clinically significant findings in laboratory tests | up to 8 days after drug administration

SECONDARY OUTCOMES:
Maximum concentration in plasma (Cmax) | up to 32 hours after first drug administration
Time to maximum concentration in plasma (tmax) | up to 32 hours after first drug administration
Terminal half-life (t1/2) | up to 32 hours after first drug administration
Area under the plasma concentration-time curve from zero to the last time points with a quantifiable plasma concentration (AUC0-tf) | up to 32 hours after first drug administration
Area under the plasma concentration-time curve extrapolated to infinity (AUC0-inf) | up to 32 hours after first drug administration
Total Mean residence time (MRTtot) | up to 32 hours after first drug administration
Total plasma clearance (CLtot) | up to 32 hours after first drug administration
Volume of distribution (Vz) | up to 32 hours after first drug administration
Volume of distribution at steady state (Vss) | up to 32 hours after first drug administration
Amount excreted into urine (Ae) | up to 32 hours after first drug administration
Mean residence time of disposition (MRTdisp) | up to 32 hours after first drug administration
Renal clearance (CLR) | up to 32 hours after first drug administration